CLINICAL TRIAL: NCT02314117
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of Capecitabine and Cisplatin With or Without Ramucirumab as First-line Therapy in Patients With Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (RAINFALL)
Brief Title: A Study of Ramucirumab (LY3009806) in Combination With Capecitabine and Cisplatin in Participants With Stomach Cancer
Acronym: RAINFALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15372; I4T-MC-JVCU (Other: Eli Lilly and Company); 2014-002240-40 (EudraCT Number)
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Ramucirumab; Capecitabine; Cisplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ramucirumab + Cisplatin + Capecitabine (Experimental): 8 milligrams/kilogram (mg/kg) ramucirumab given intravenously (IV) on days 1 and 8 in combination with 80 mg/square meter (m^2) cisplatin given IV on day 1 of each 21-day cycle (for up to 6 cycles) and 1000 mg/m^2 capecitabine given orally twice a day on days 1 through 14. Participants that were unable to take capecitabine will be given 800 mg/m^2/day fluorouracil (5-FU) IV on days 1 to 5 of each 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Capecitabine; Drug: Cisplatin; Drug: Fluorouracil
- Placebo + Cisplatin + Capecitabine (Active Comparator): Placebo for blinding given IV on days 1 and 8 in combination with 80 mg/m^2 cisplatin given IV on day 1 of each 21-day cycle (for up to 6 cycles) and 1000 mg/m^2 capecitabine given orally twice a day on days 1 through 14. Participants that were unable to take capecitabine will be given 800 mg/m^2/day 5-FU IV on days 1 to 5 of each 21-day cycle.
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Placebo; Drug: Fluorouracil

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B; Cyramza
  Arms: Ramucirumab + Cisplatin + Capecitabine
Drug: Capecitabine — Administered orally
Drug: Cisplatin — Administered IV
Drug: Placebo — Administered IV
  Arms: Placebo + Cisplatin + Capecitabine
Drug: Fluorouracil — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the efficacy of ramucirumab, which is a targeted antibody, in combination with capecitabine and cisplatin compared to capecitabine and cisplatin alone in participants with stomach cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a histopathologically confirmed diagnosis of metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma. All histologies of nonsquamous cell origin including undifferentiated gastric carcinoma are eligible.
* Have not received any prior first-line systemic therapy (prior adjuvant or neo-adjuvant therapy is permitted). Participants whose disease has progressed after >12 months following the last dose of systemic treatment in the adjuvant/neoadjuvant setting are eligible.
* Have measurable or nonmeasurable but evaluable disease determined using guidelines in Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v 1.1). Baseline tumor assessment should be performed using a high resolution computed tomography (CT) scan using IV and oral contrast unless clinically contra-indicated. Magnetic resonance imaging (MRI) is acceptable if a CT cannot be performed.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group scale at baseline.
* Have adequate organ function.
* Have baseline clinical and laboratory parameters that are consistent with the requirements prescribed in respective labels and are suitable for consideration of treatment with capecitabine (or 5-FU) and cisplatin (for example, dihydropyrimidine dehydrogenase deficiency).
* Have an estimated life expectancy of ≥12 weeks in the judgment of the investigator.

Exclusion Criteria:

* Participants with adenocarcinoma of the esophagus are excluded.
* Participants with human epidermal growth factor receptor 2 (HER2)-positive status.
* Participants receiving chronic therapy with nonsteroidal anti-inflammatory agents.
* Have radiation therapy within 14 days prior to randomization.
* Have documented brain metastases, leptomeningeal disease or uncontrolled spinal cord compression.
* Have significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal tract within 12 weeks prior to randomization.
* Have experienced any arterial thromboembolic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization.
* Have symptomatic congestive heart failure (New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
* Have uncontrolled hypertension prior to initiating study treatment, despite antihypertensive intervention.
* Have undergone major surgery within 28 days prior to randomization, or central venous access device placement within 7 days prior to first dose of study treatment, except if the procedure is minimally invasive (for example, introduction of peripherally inserted central catheter [PICC] line) and the investigator does not anticipate any significant bleeding.
* Have a history of gastrointestinal perforation and/or fistulae within 6 months prior to randomization.
* Have a history of inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to randomization.
* Have an acute or subacute bowel obstruction or history of chronic diarrhea which is considered clinically significant in the opinion of the investigator.
* The participant has:

  * cirrhosis at a level of Child-Pugh B (or worse) or
  * cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
* Have known allergy or hypersensitivity to any components of study treatment.
* Are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (125):
- United States (25):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St Jude Medical Center, Fullerton, California
  - SMO TRIO -Translational Research, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology Corporation, Santa Monica, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - Illinois CancerCare, Peoria, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - UT Southwestern Med Ctr, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Argentina (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viedma, Río Negro Province
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario, Santa Fe Province
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rioja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salta
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vancouver
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hradec Králové
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olomouc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus C
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense C
- Finland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avignon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clermont-Ferrand
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt am Main
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaposvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- Israel (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Italy (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrette Di Ancona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
- Japan (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Higashinari-Ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kashiwa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitaadachi-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kōtoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suita-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunto-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utsunomiya
- Mexico (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara, Jalisco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Bernardino, Toluca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juchitán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., México
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oaxaca City
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nieuwegein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sittard - Geleen
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (4):
  - Ad-Vance Medical Research, Ponce
  - Hospital Espanol Auxilio Mutuo, San Juan
  - VA Caribbean Healthcare System, San Juan
  - Hospital Municipal de San Juan, San Juan
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elche
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
- United Kingdom (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merseyside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Fuchs CS, Shitara K, Di Bartolomeo M, Lonardi S, Al-Batran SE, Van Cutsem E, Ilson DH, Alsina M, Chau I, Lacy J, Ducreux M, Mendez GA, Alavez AM, Takahari D, Mansoor W, Enzinger PC, Gorbounova V, Wainberg ZA, Hegewisch-Becker S, Ferry D, Lin J, Carlesi R, Das M, Shah MA; RAINFALL Study Group. Ramucirumab with cisplatin and fluoropyrimidine as first-line therapy in patients with metastatic gastric or junctional adenocarcinoma (RAINFALL): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):420-435. doi: 10.1016/S1470-2045(18)30791-5. Epub 2019 Feb 1. PMID 30718072
- See also: A Study of Ramucirumab (LY3009806) in Combination With Capecitabine and Cisplatin in Participants With Stomach Cancer — https://trials.lillytrialguide.com/en-US/trial/kPN4NxC5uCCu4eG6MMGeI?conditionId=B6nAiYh98OCsos8uoOISQ

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as participants who died or those who were alive and off treatment when the study completed.
Period: Overall Study
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Started | 326 | 319
Received at Least One Dose of Study Drug | 323 | 315
Completed | 314 | 303
Not Completed | 12 | 16
Not completed — Lost to Follow-up | 9 | 14
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine | Total
Number analyzed (Participants) | 326 | 319 | 645
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (11.6) | 60.1 (11.8) | 59.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 104 | 216
  Male | 214 | 215 | 429
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 62 | 129
  Not Hispanic or Latino | 227 | 245 | 472
  Unknown or Not Reported | 32 | 12 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 11 | 23
  Asian | 38 | 31 | 69
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 256 | 264 | 520
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 10 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 1 | 1 | 2
  Argentina | 21 | 22 | 43
  Hungary | 15 | 16 | 31
  United States | 42 | 31 | 73
  Czechia | 11 | 8 | 19
  Japan | 32 | 28 | 60
  United Kingdom | 20 | 22 | 42
  Russia | 25 | 25 | 50
  Spain | 10 | 13 | 23
  Canada | 10 | 6 | 16
  Netherlands | 4 | 7 | 11
  Belgium | 8 | 5 | 13
  Finland | 3 | 5 | 8
  Denmark | 12 | 3 | 15
  Poland | 8 | 10 | 18
  Italy | 28 | 45 | 73
  Mexico | 26 | 26 | 52
  Israel | 11 | 12 | 23
  France | 19 | 21 | 40
  Germany | 20 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS time was measured from the date of randomization to the date of radiographic(rgr) documentation of progression(by RECIST v.1.1) or the date of death due to any cause, whichever was earlier.If a participant did not have a complete baseline tumor assessment,then the PFS time was censored at the randomization date.If a participant was not known to have died or have rgr documented progression as of the data cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date. If death or progressive disease(PD) occurred after 2 or more consecutive missing rgr visits,censoring occurred at the date of the last rgr visit prior to the missed visits.If death or PD occurred after postdiscontinuation(pdis) systemic anticancer therapy,censoring occurred at the date of last rgr visit prior to the start of pdis systemic anticancer therapy. PD was defined according to RECIST v.1.1.
Time Frame: Randomization to Radiological Disease Progression or Death from Any Cause (Up to 26 Months)
Population: First 508 randomized participants. Participants censored: Ramucirumab + Cisplatin + Capecitabine=87 and Placebo + Cisplatin + Capecitabine=62.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 255 | 253
months | 5.72 [5.45 to 6.51] | 5.39 [4.47 to 5.72]
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 0.753, 95% CI 2-sided [0.607 to 0.935]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was time from the date of randomization to the date of death from any cause. If the participant was alive at the cutoff for analysis (or was lost to follow-up), OS data were censored for analysis on the last date the participant was known to be alive.
Time Frame: Randomization to Death from Any Cause (Up To 30 Months)
Population: All randomized participants. Participants censored: Ramucirumab + Cisplatin + Capecitabine=87 and Placebo + Cisplatin + Capecitabine=88.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
months | 11.17 [9.92 to 11.93] | 10.74 [9.53 to 11.89]
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 0.962, 95% CI 2-sided [0.801 to 1.156]

3. Secondary Outcome: Progression- Free Survival 2 (PFS2)
Description: PFS2 was defined as the time from the date of randomization to second disease progression (defined as objective radiological or symptomatic progression), or death of any cause, whichever occurs first. Participants alive and for whom a second disease progression has not been observed (including participants who did not receive any additional systemic anticancer treatments) were censored at the last time known to be alive and without second disease progression. The second progression refers to disease progression on or after additional systemic anticancer therapy, regardless if any earlier progression is observed or not(e.g. at the end of study treatment). It is assessed by investigator based on overall clinical evaluation, not limited to RECIST.
Time Frame: Randomization to Second Radiological or Symptomatic Disease Progression After the Start of Additional Systemic Anticancer Treatment or Death from Any Cause (Up To 26 Months)
Population: All randomized participants. Participants censored: Ramucirumab + Cisplatin + Capecitabine=74 and Placebo + Cisplatin + Capecitabine=74.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
months | 10.18 [9.03 to 10.84] | 9.20 [8.34 to 9.99]
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 0.926, 95% CI 2-sided [0.774 to 1.108]

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1).Target lesions - CR: Disappearance of all lesions; any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of lesions vs the baseline sum. PD: At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study (the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s). Non target lesions - CR: Disappearance of all lesions and normalization of tumor marker levels; all lymph nodes must be non-pathological in size. Non-CR/Non-PD: Persistence of lesion(s) and/or maintenance of abnormal tumor marker levels. PD: Unequivocal progression of existing lesions or the appearance of new lesion(s).ORR calculated as:(sum of the number of participants with PRs and CRs) divided by (number of evaluable participants) multiplied by 100.
Time Frame: Randomization to Disease Progression (Up To 26 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
percentage of participants | 41.1 [35.8 to 46.4] | 36.4 [31.1 to 41.6]

5. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD) (Disease Control Rate [DCR])
Description: DCR was the percentage of participants with a best overall response of CR, PR, or SD as per Response using RECIST v1.1 criteria. Target lesions - CR: Disappearance of all lesions; any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of lesions vs the baseline sum. Progressive Disease (PD): At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study (the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s). Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Non target lesions - CR: Disappearance of all lesions and normalization of tumor marker levels; all lymph nodes must be non-pathological in size. Non-CR/Non-PD: Persistence of lesion(s) and/or maintenance of abnormal tumor marker levels. PD: Unequivocal progression of existing lesions or the appearance of new lesion(s).
Time Frame: Randomization to Disease Progression (Up To 26 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo + Cisplatin + Capecitabine: Placebo for blinding given IV on days 1 and 8 in combination with 80 mg/m^2 cisplatin given IV on day 1 of each 21 day cycle (for up to 6 cycles) and 1000 mg/m^2 capecitabine given orally twice a day on days 1 through 14. Participants that are unable to take capecitabine will be given 800 mg/m^2/day 5-FU IV on days 1 to 5 of each 21 day cycle.
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
percentage of participants | 81.9 [77.7 to 86.1] | 76.5 [71.8 to 81.1]

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP was time from the date of randomization to the date of radiographic progression (according to RECIST v.1.1). If a participant died due to any reason without radiographic progression, TTP is censored at the last adequate tumor assessment. Target lesions: Progressive Disease (PD): At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study (the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s). Non target lesions: PD: Unequivocal progression of existing lesions or the appearance of new lesion(s).
Time Frame: Randomization to Disease Progression (Up To 24 Months)
Population: All randomized participants. Participants censored: Ramucirumab + Cisplatin + Capecitabine=149 and Placebo + Cisplatin + Capecitabine=111.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
months | 6.77 [5.88 to 7.66] | 5.78 [5.55 to 6.37]
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 0.699, 95% CI 2-sided [0.569 to 0.859]

7. Secondary Outcome: Duration of Response (DoR)
Description: Participants achieved an objective response if they had a best overall response of CR or PR.Target lesions- CR:Disappearance of all lesions;any pathological lymph nodes must have reduction in short axis to <10 mm.PR: At least a 30% decrease in the sum of diameters of lesions vs the baseline sum.PD: At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study(the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s).Non target lesions - CR: Disappearance of all lesions and normalization of tumour marker levels;all lymph nodes must be non-pathological in size. Non-CR/Non-PD:Persistence of lesion(s) and/or maintenance of abnormal tumor marker levels.PD:Unequivocal progression of existing lesions or the appearance of new lesion(s).If a participant was not known to have died or have radiographically documented PD as of the data inclusion cutoff date,DOR was censored at the date of the last adequate tumor assessment.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up To 26 Months)
Population: All randomized participants. Participants censored : Ramucirumab + Cisplatin + Capecitabine= 23 and Placebo + Cisplatin + Capecitabine=10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 134 | 116
months | 5.72 [5.09 to 6.34] | 4.27 [3.88 to 4.90]
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.499 to 0.866]

8. Secondary Outcome: Time to Deterioration in Quality of Life (QoL) on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) - Global Health Status/ QoL Scale
Description: Time to sustained deterioration was defined as time from randomization to first worsening in QoL with no subsequent non-worsened assessment. Worsening in global health status/QoL was defined as a decrease of ≥10 points on a 100-point scale. If a participant did not report worsening, time to sustained deterioration was censored at date of last non-worsened assessment.
Time Frame: Randomization, First worsening in QoL (Up To 26 Months)
Population: All randomized participants. Participants censored: Ramucirumab + Cisplatin + Capecitabine=215 and Placebo + Cisplatin + Capecitabine=217
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
months | 9.00 [8.08 to 12.58] | 9.46 [6.74 to 11.99]
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 1.013, 95% CI 2-sided [0.770 to 1.332]

9. Secondary Outcome: Change in Health Status on the EuroQol 5-Dimensions 5-Level Instrument (EQ-5D- 5L)
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Five dimensions of health status are each assessed with 5 response options and scored as a composite index which were anchored on a scale of 0 to 1 with a higher score representing better health status. Additionally, current health status was assessed on a visual analogue scale (VAS) ranging from 0 to 100 with a higher score representing better health status.
Time Frame: Randomization, 30 Days After Treatment Discontinuation (Up To 5 Months)
Population: All randomized participants who provided data at baseline and cycle 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 136 | 125
units on a scale
  EQ-5D index | -0.008 (0.148) | -0.010 (0.157)
  EQ-5D VAS | 0.8 (18.56) | 1.5 (20.33)

10. Secondary Outcome: Time to Deterioration in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: The time from the date of randomization to the first date observing ECOG PS ≥2 (that is, deterioration from baseline status of 0 or 1). Participants without PS deterioration were censored at their last documented assessments of 0 or 1. ECOG Performance Status: 2- Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours, 3 -Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours, 4 -Completely disabled. Cannot carry on any selfcare.Totally confined to bed or chair,5- Dead.
Time Frame: Randomization to ECOG PS ≥2 (Up To 26 Months)
Population: All randomized participants. Participants censored: Ramucirumab + Cisplatin + Capecitabine=254 and Placebo + Cisplatin + Capecitabine= 260.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 326 | 319
months | NA [12.2 to NA] — Very few events occurred therefore data were not assessable. | NA [NA to NA] — Very few events occurred therefore data were not assessable.
Statistical Analysis 1: Comparison: Ramucirumab + Cisplatin + Capecitabine vs Placebo + Cisplatin + Capecitabine; Test type: Superiority; Hazard Ratio (HR) = 1.117, 95% CI 2-sided [0.790 to 1.580]

11. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: Participants who developed treatment-emergent antibody responses to Ramucirumab postbaseline.
Time Frame: Predose Cycle 1 through 30 Days After Treatment Discontinuation (Up To 24 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Cisplatin + Capecitabine | Placebo + Cisplatin + Capecitabine
Number analyzed (Participants) | 323 | 315
Participants | 4 | 5

12. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Ramucirumab
Description: Pharmacokinetics (PK): Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Ramucirumab
Time Frame: Cycle 1 Day 1: 1 hour (hr) end of infusion (EOI), Cycle 3 Day 1: 1hr EOI, Cycle 9 Day 1: 1 hr EOI
Population: All randomized participants who received ramucirumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter (µg/mL)
Arm/Group | Ramucirumab + Cisplatin + Capecitabine
Number analyzed (Participants) | 283
Microgram/milliliter (µg/mL)
  Cycle 1, Day 1 | 133 (31)
  Cycle 3, Day 1: number analyzed (Participants) | 146
  Cycle 3, Day 1 | 173 (35)
  Cycle 9, Day 1: number analyzed (Participants) | 16
  Cycle 9, Day 1 | 169 (60)

13. Secondary Outcome: PK: Minimum Concentration (Cmin) of Ramucirumab
Description: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Time Frame: Cycle 1 Day 1: 1 hour (hr) end of infusion (EOI), Cycle 3 Day 1: 1hr EOI, Cycle 9 Day 1: 1 hr EOI
Population: All randomized participants who received ramucirumab and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab + Cisplatin + Capecitabine
Number analyzed (Participants) | 268
µg/mL
  Cycle 1, Day 8 | 40.7 (35)
  Cycle 2, Day 1: number analyzed (Participants) | 232
  Cycle 2, Day 1 | 35.7 (56)
  Cycle 3, Day 1: number analyzed (Participants) | 163
  Cycle 3, Day 1 | 51.2 (47)
  Cycle 5, Day 1: number analyzed (Participants) | 85
  Cycle 5, Day 1 | 69.7 (52)
  Cycle 9, Day 1: number analyzed (Participants) | 21
  Cycle 9, Day 1 | 77.6 (98)

ADVERSE EVENTS:
Time Frame: Baseline Up To 5.6 Years
Description: All participants who received at least one dose of study drug.
Groups:
- LY3009806+Capecitabine+Cisplatin: 8 milligrams/kilogram (mg/kg) ramucirumab given intravenously (IV) on days 1 and 8 in combination with 80 mg/square meter (m^2) cisplatin given IV on day 1 of each 21-day cycle (for up to 6 cycles) and 1000 mg/m^2 capecitabine given orally twice a day on days 1 through 14. Participants that were unable to take capecitabine will be given 800 mg/m^2/day fluorouracil (5-FU) IV on days 1 to 5 of each 21-day cycle.
- Placebo+Capecitabine+Cisplatin: Placebo for blinding given IV on days 1 and 8 in combination with 80 mg/m^2 cisplatin given IV on day 1 of each 21-day cycle (for up to 6 cycles) and 1000 mg/m^2 capecitabine given orally twice a day on days 1 through 14. Participants that were unable to take capecitabine will be given 800 mg/m^2/day 5-FU IV on days 1 to 5 of each 21-day cycle.
Arm/Group | LY3009806+Capecitabine+Cisplatin | Placebo+Capecitabine+Cisplatin
Serious Adverse Events (participants affected / at risk) | 161/323 | 150/315
Other Adverse Events (participants affected / at risk) | 315/323 | 304/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3009806+Capecitabine+Cisplatin (N=323) | Placebo+Capecitabine+Cisplatin (N=315)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 11 (16)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 11 (13)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 8 (9)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (16) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 19 (20)
Dysphagia (Gastrointestinal disorders) | 8 (9) | 7 (8)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 5 (5) | 3 (3)
Gastric perforation (Gastrointestinal disorders) | 9 (9) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (3) | 3 (5)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 4 (7) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 8 (10)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Subileus (Gastrointestinal disorders) | 4 (5) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5) | 1 (2)
Vomiting (Gastrointestinal disorders) | 14 (15) | 22 (27)
Asthenia (General disorders) | 3 (3) | 2 (2)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 2 (2)
Fall (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 6 (7) | 5 (5)
Heparin-induced thrombocytopenia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (4) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 3 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 2 (2) | 12 (12)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (2)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 4 (5) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 7 (9) | 9 (9)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 10 (10) | 8 (13)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 3 (3)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis deep (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3009806+Capecitabine+Cisplatin (N=323) | Placebo+Capecitabine+Cisplatin (N=315)
Anaemia (Blood and lymphatic system disorders) | 104 (276) | 114 (289)
Neutropenia (Blood and lymphatic system disorders) | 71 (218) | 74 (133)
Thrombocytopenia (Blood and lymphatic system disorders) | 41 (106) | 26 (51)
Tinnitus (Ear and labyrinth disorders) | 23 (26) | 27 (32)
Abdominal pain (Gastrointestinal disorders) | 52 (80) | 51 (69)
Abdominal pain upper (Gastrointestinal disorders) | 22 (27) | 15 (22)
Constipation (Gastrointestinal disorders) | 104 (161) | 78 (107)
Diarrhoea (Gastrointestinal disorders) | 108 (175) | 107 (175)
Dyspepsia (Gastrointestinal disorders) | 19 (20) | 12 (14)
Dysphagia (Gastrointestinal disorders) | 21 (33) | 17 (23)
Nausea (Gastrointestinal disorders) | 205 (459) | 186 (444)
Stomatitis (Gastrointestinal disorders) | 67 (110) | 39 (64)
Vomiting (Gastrointestinal disorders) | 134 (249) | 117 (217)
Asthenia (General disorders) | 44 (133) | 40 (101)
Fatigue (General disorders) | 153 (316) | 145 (309)
Mucosal inflammation (General disorders) | 20 (31) | 17 (41)
Oedema peripheral (General disorders) | 45 (65) | 33 (46)
Pyrexia (General disorders) | 28 (37) | 40 (56)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 17 (18)
Alanine aminotransferase increased (Investigations) | 19 (29) | 10 (15)
Aspartate aminotransferase increased (Investigations) | 20 (25) | 12 (17)
Blood creatinine increased (Investigations) | 31 (60) | 28 (41)
Neutrophil count decreased (Investigations) | 103 (295) | 92 (263)
Platelet count decreased (Investigations) | 72 (254) | 33 (75)
Weight decreased (Investigations) | 54 (72) | 37 (56)
White blood cell count decreased (Investigations) | 37 (118) | 32 (109)
Decreased appetite (Metabolism and nutrition disorders) | 130 (245) | 100 (190)
Dehydration (Metabolism and nutrition disorders) | 19 (25) | 25 (30)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (28) | 13 (21)
Hypocalcaemia (Metabolism and nutrition disorders) | 20 (23) | 11 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 36 (51) | 40 (68)
Hypomagnesaemia (Metabolism and nutrition disorders) | 36 (47) | 45 (97)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (30) | 17 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (33) | 16 (20)
Dizziness (Nervous system disorders) | 36 (42) | 35 (52)
Dysgeusia (Nervous system disorders) | 34 (38) | 27 (31)
Headache (Nervous system disorders) | 43 (57) | 27 (36)
Neuropathy peripheral (Nervous system disorders) | 20 (30) | 8 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 39 (62) | 31 (41)
Insomnia (Psychiatric disorders) | 27 (29) | 25 (27)
Proteinuria (Renal and urinary disorders) | 64 (156) | 36 (60)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 18 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 (49) | 21 (26)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48 (76) | 14 (19)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 36 (63) | 33 (46)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (21) | 16 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (23) | 16 (17)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 99 (248) | 63 (121)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 18 (18) | 10 (10)
Embolism venous (Vascular disorders) | 13 (13) | 17 (17)
Hypertension (Vascular disorders) | 70 (152) | 23 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days